CLINICAL TRIAL: NCT00343109
Title: Phase II Study of a HER-2/Neu (HER2) Intracellular Domain (ICD) Peptide-Based Vaccine Administered to Patients With Locally Advanced or Stage IV HER2 Positive Breast Cancer
Brief Title: Vaccine Therapy in Treating Patients Receiving Trastuzumab For HER2-Positive Stage IIIB-IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6166 (FH/UWCC ID); NCI-2010-00803 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BC 030289 (Other: Department of Defense Breast Cancer Program); 120 (Other: Tumor Vaccine Group); NCT00369525 (obsolete NCT alias)
Record Dates: First submitted 2006-06-20; First posted 2006-06-22 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2019-05

CONDITIONS: HER2-positive Breast Cancer; Male Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Leukapheresis; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Immunologic Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): Patients receive HER-2/neu intracellular domain peptide-based vaccine mixed with GM-CSF intradermally once monthly for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: HER-2/neu intracellular domain protein; Procedure: leukapheresis; Other: laboratory biomarker analysis; Biological: sargramostim; Other: immunologic technique; Biological: synthetic tumor-associated peptide vaccine therapy

INTERVENTIONS:
Biological: HER-2/neu intracellular domain protein — Given ID
  Other Names: HER-2 ICD Peptide; HER-2/neu ICD Protein
Procedure: leukapheresis — Optional correlative studies
Other: laboratory biomarker analysis — Correlative studies
Biological: sargramostim — Given ID
  Other Names: GM-CSF; Leukine; Prokine
Other: immunologic technique — Correlative studies
  Other Names: immunological laboratory methods; laboratory methods, immunological
Biological: synthetic tumor-associated peptide vaccine therapy — Given ID

SUMMARY:
This phase II trial is studying how well vaccine therapy works in treating patients receiving trastuzumab for HER2-positive stage IIIB- IV breast cancer. Vaccines made from peptides may help the body build an effective immune response to kill tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To estimate the RFS in patients with HER2 positive locally advanced breast cancer vaccinated with a HER2 ICD peptide-based vaccine.

SECONDARY OBJECTIVES:

1. To assess the safety of a HER2 ICD peptide-based vaccine administered concurrently with trastuzumab.
2. To determine the immunogenicity of the HER2 ICD peptide based vaccine when given within one year of initiating standard treatment which includes trastuzumab.

   1. To determine the incidence of the development of T cell immunity specific for the HER2 ICD.
   2. To determine the incidence of the development of intramolecular epitope spreading.
   3. To determine the magnitude of the HER2 ICD specific CD4+ and CD8+ immune response generated with immunization.
3. To assess whether there is an association between RFS and the development of an immune response (HER2 specific T cell immunity and/or the development of intramolecular epitope spreading).

OUTLINE:

Patients receive HER-2/neu intracellular domain peptide-based vaccine mixed with GM-CSF intradermally (ID) once monthly for 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1, 4, 8, and 12 months and then annually thereafter for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB or Stage IIIC breast cancer who are within 1 year of diagnosis and initiating treatment with chemotherapy and trastuzumab; and are in complete remission
* Stage IV breast cancer in first complete remission and defined as NED (no evidence of disease) or with stable bone only disease who are within 6 months of initiating maintenance trastuzumab
* NED status should be documented by chest/abdominal CT, PET or PET/CT within the last 90 days
* Bone only disease documented as stable or healed by PET, PET/CT, or MRI within the last 90 days; stable bone-only disease must be documented with bone scan performed within the last 6 months
* HER2 overexpression by IHC of 2+ or 3+, in the primary tumor or metastasis or documented gene amplification by FISH analysis; if overexpression is 2+ by IHC, then patients must have HER2 gene amplification documented by FISH
* Eligible subjects must have been treated to NED or stable bone only disease status with trastuzumab and/or chemotherapy and be off cytotoxic chemotherapy or immunosuppressive agents (e.g. systemic steroids) for at least 30 days prior to enrollment (concurrent hormonal therapy allowed; concurrent bisphosphonate therapy allowed)
* Patients on trastuzumab should continue trastuzumab monotherapy per standard of care (the dosing and schedule of trastuzumab should follow standard guidelines as described below: trastuzumab 2mg/kg IV weekly or trastuzumab 6mg/kg IV every 3 weeks)
* Subjects must have an ECOG Performance Status Score =< 1
* Non-menopausal female subjects must agree to contraception for the remainder of their childbearing years
* Male subjects must use an acceptable form of contraception throughout the course of the study
* Hematocrit >= 30,000
* Platelet count >= 100,000
* WBC >= 3000/mcl
* Stable creatinine =< 2.0 mg/dl or a creatinine clearance greater than 60 ml/min
* Serum bilirubin < 1.5 mg/dl
* SGOT < 2x ULN
* Laboratory tests should be performed within 60 days of enrollment
* Subjects must have recovered from major infections and/or surgical procedures and, in the opinion of the investigator, not have any significant active concurrent medical illnesses precluding protocol treatment
* Patients on trastuzumab monotherapy must have adequate cardiac function as demonstrated by normal ejection fraction (EF) on MUGA scan or echocardiogram performed within last 6 months

Exclusion Criteria:

* Subjects cannot be simultaneously enrolled in other treatment studies
* Patients cannot be receiving any other concurrent immunomodulators besides trastuzumab
* Any contraindication to receiving GM-CSF based vaccine products
* Cardiac disease, specifically restrictive cardiomyopathy, unstable angina within the last 6 months prior to enrollment, New York Heart Association functional class III-IV heart failure on active treatment with normalized LVEF on therapy, and symptomatic pericardial effusion
* Active autoimmune disease
* Subjects can not have active immunodeficiency disorder, e.g. HIV
* Cannot be pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-03; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival | At 4 years

SECONDARY OUTCOMES:
Safety as assessed by NCI CTCAE version 3.0 | Baseline and 1 month following last vaccination
Immune response as assessed by HER2 specific T cell immunity and/or intramolecular epitope spreading | Baseline, midpoint in the immunization schedule (prior to the 4th vaccine), 1 month after the 6th and last immunization and at 4, 8 and 12 months after the end of vaccinations
Correlation of RFS to the generation of an immune response | Prior to the 4th vaccine, 1 month after the 6th and last immunization and at 4, 8 and 12 months after the end of vaccinations

CONTACTS AND LOCATIONS:
Overall Officials: Mary Disis, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States